CLINICAL TRIAL: NCT03727633
Title: Traitement Des Carcinomes hépatocellulaires Sur Cirrhose Child A/B7 Par Injection Intra-artérielle hépatique d'Une émulsion de Lipiodol et Idarubicine : Etude de Phase II, Monobras, Multicentrique.
Brief Title: Hepatocellular Carcinoma on Cirrhosis With Child A/B7 and Hepatic Intra Arterial Injection of Idarubicin/Lipiodol Emulsion
Acronym: LIDA-BII
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: University Hospital, Montpellier (Other)
Collaborators: Guerbet (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RECHMPL17_0304; 2017-004859-22 (EudraCT Number); UF 9888 (Other: Montpellier University Hospital)
Record Dates: First submitted 2018-05-31; First posted 2018-11-01 (Actual); Last update posted 2026-01-05 (Actual); Status verified 2025-12

CONDITIONS: Carcinoma, Hepatocellular
MeSH Terms: conditions — Carcinoma, Hepatocellular | interventions — Idarubicin; Ethiodized Oil

STUDY DESIGN:
Intervention Model Description: The purpose of this study is to assess efficacy and tolerance of hepatic intra-arterial injection of an emulsion of Idarubicine and Lipiodol for treatment of non-metastatic, unresectable hepatocellular carcinoma on cirrhosis with Child-Pugh A/B7.
Masking Description: No masking is used. All involved know the identity of the intervention assignment.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Treatment arm (Experimental): hepatic intra-arterial injection of an emulsion of Idarubicine and Lipiodol
  Interventions: Drug: Idarubicin and Lipiodol

INTERVENTIONS:
Drug: Idarubicin and Lipiodol — Hepatic intra-arterial chemotherapy consisting of the hepatic intra-arterial injection Idarubicin, emulsified with Lipiodol

SUMMARY:
The investigators propose in this trial to test a hepatic chemotherapy, consisting of the hepatic intra-arterial injection Idarubicin, emulsified with Lipiodol, lipid vector, without embolization in the treatment of non-metastatic, unresectable hepatocellular carcinoma on cirrhosis with Child-Pugh A/B7.

ELIGIBILITY:
Inclusion Criteria:

* Histologically-proven HCC or according to EASL criteria
* Child-Pugh A or B7
* Disease that is not suitable for resection, ablation or radiofrequency
* Performance Status ECOG 0 or 1
* BCLC A/B or C if Performance Status ECOG = 1
* Measurable lesions according to mRECIST criteria
* No previous treatment with chemotherapy, radiotherapy or transarterial embolization (with or without chemotherapy) or radioembolisation
* Age superior or equal to 18 years
* Platelets > 50,000/mm3, Polynuclear neutrophils > 1000/mm3, Creatininemia < 150umol/L, Bilirubinemia < 5 mg/dL
* Absence of heart failure (Ultrasound LVEF > 50%)
* Women of child-bearing age using an adequate method of contraception throughout treatment
* Men using an adequate method of contraception throughout the treatment and at least 3 months after the end of treatment
* Written informed consent
* National health insurance cover

Exclusion Criteria:

* Advanced tumor disease (extrahepatic except pulmonary micronodules <7mm of tumoral portal vein thrombosis on positron emission tomography are not a contra-indication.)
* Large HCC with liver invasion >50%
* History of other cancer than HCC and excluding cancers known to have been cured for more than 5 years, or basocellular skin tumors or cervical cancer in situ treated with adequate and curative purpose
* Advanced liver disease (Child B8, B9 or C)
* Contra-indication for the MRI (Pacemaker or neurosensorial stimulator or implantable defibrillator, cochlear implant, ferromagnetic foreing body similar to the nervous structure)
* Contra-indication to the injection of the gadolinium-based contrast agents (history of hypersensibility to the gadolinium chelates, meglumine).
* Contra-indication to idarubicin (Hypersensibility to active substance or excipients, cardiopathy with myocardial insufficiency of less than 6 months, serious arrhythmias, serious renal or liver failure, yellow fever vaccine or any other live attenuated vaccine, persistente myelosuppression, previous treatments with idarubicin and/or other anthracyclines or anthracenediones at maximum cumulative doses, stomatitis)
* Contra-indication to Lipiodol (Hypersensibility, proven hyperthyroidism, tromatic injuries, bleeding or recent bleeding)
* Concomitant disease or uncontrolled severe clinical situation
* Uncontrolled severe infection
* Vascular anatomy makes it impossible to perform hepatic intra-arterial treatments
* Pregnancy (Beta HCG positive) or breastfeeding
* Patient who for psychological, social, family or geographical reasons cannot be followed regularly
* Vulnerable person
* Concomitant participation of the patient in another research involving the human person

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 53 (Estimated)
Dates: Start 2018-07-19 (Actual); Primary Completion 2025-06-18 (Actual); Study Completion 2026-06-18 (Estimated)

PRIMARY OUTCOMES:
Percentage of participants presenting a disease control at 4 months | 4 months
  The primary outcome is to evaluate the disease control rate (partial, complete or stable response) 4 months after the first cycle of chemo-lipiodol using mRECIST criteria.

SECONDARY OUTCOMES:
Safety of chemo-lipiodol defined by NCI-CTCAE version 4.03 | 12 months
  Safety defined by NCI-CTCAE version 4.03 published 14 june 2010
Objective response rate of chemo-lipiodol | 6 months
  Objective response rate according to mRECIST at 6 months after the first cycle
best response at 6 months after the first cycle of chemo-lipiodol according to mRECIST | 6 months
  The best response according to mRECIST at 6 months after the first cycle of chemo-lipiodol
Overall survival | 12 months
  Overall survival at 12 months after the first cycle of chemo-lipiodol
Quality of life questionnaire (QLQ) QLQ-C30 | 12 months
  Quality of life questionnaire at 12 months after the first cycle of chemo-lipiodol (QLQ-C30). Subscale minimum score is egal to 1 (not at all) and maximum score is egal to 4 (very much). The maximal score correspond to a better quality of life. Subscales are summed to compute a total score.

CONTACTS AND LOCATIONS:
Overall Officials: Boris GUIU, Principal Investigator — Montpellier University Hospital
Locations (4):
- France (4):
  - CHU d'Angers, Angers
  - CHU de Dijon, Dijon
  - CHU de Montpellier, Montpellier
  - CHU de Nice, Nice